CLINICAL TRIAL: NCT05725863
Title: The Effect of Mindfulness-Based Cognitive Therapy Applied to Postpartum Mothers on Stress, Postpartum Blues, Mother-Baby Attachment and Breastfeeding
Brief Title: Mindfulness-Based Cognitive Therapy Postpartum Mothers Stress, Postpartum Blues, Mother-Baby Attachment and Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Principal Investigator, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/P004
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Mindfulness-based Cognitive Therapy
Keywords: Postpartum; Stress; Postpartum blues; Mother-infant attachment; Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No psychological intervention was offered. Postpartum mothers in the control condition were informed that they would receive MBCT after a waiting period of 2 months.
- MBCT (Experimental): Mindfulness-Based Cognitive Therapy (MBCT) consisted of eight weekly 2.5-hr sessions and one 3-hr silent session. First, psycho-education focused on the importance of recognizing personal feelings and the relationship between stress, postpartum blues, mother-infant attachment and breastfeeding symptoms, and stress management, stress, postpartum blues, mother-infant attachment and breastfeeding. Additionally, postpartum mothers' experiences of stress, postpartum blues, mother-infant attachment, and breastfeeding were central during the study and were a recurring topic for the purpose of the study in general. Postpartum mothers were given homework assignments, including audio CDs with formal exercises, and were asked to practice for 30 min per day.
  Interventions: Other: Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Other: Mindfulness-Based Cognitive Therapy — Mindfulness-Based Cognitive Therapy (MBCT) is a structured group intervention developed by Segal et al. (2002). The intervention consisted of eight weekly 2.5-hr sessions and one 3-hr silent session. First, psycho-education focused on the importance of recognizing personal feelings and the relationship between stress, postpartum blues, mother-infant attachment and breastfeeding symptoms, and stress management, stress, postpartum blues, mother-infant attachment and breastfeeding. Additionally, postpartum mothers' experiences of stress, postpartum blues, mother-infant attachment, and breastfeeding were central during the study and were a recurring topic for the purpose of the study in general. Postpartum mothers were given homework assignments, including audio CDs with formal exercises, and were asked to practice for 30 min per day.
  Arms: MBCT

SUMMARY:
Objectives: Research on the effect of mindfulness-based cognitive therapy (MBCT) applied to postpartum mothers on the mother's mood and mother-infant interaction is a new and promising feld of research. However, the evidence on whether MBCT reduces stress and postpartum blues and improves mother-infant attachment and breastfeeding is inconclusive. The present study addresses this research question.

Design: A two-arm randomized controlled trial was conducted in 90 postpartum mothers.

DETAILED DESCRIPTION:
This two-arm randomized controlled trial (RCT) was conducted in the postpartum mothers located in Edirne, between April and December 2022. During the intake, postpartum mothers were informed about the goals and setup of the study and intervention, and assessed for eligibility by a brief standardized interview. Postpartum mothers who fulfilled our criteria received an information letter and informed consent form, as well as the baseline questionnaire. Those postpartum mothers that provided written informed consent for participation were included in the study. Assessments in both groups were performed before randomization (i.e., baseline) and directly after the intervention period (i.e., post-measurement, approximately 2 months after baseline).

Randomization: Postpartum mothers were randomly assigned to an 8-week MBCT or control condition. A research assistant not actively involved in the design and data analysis of the study created a random distribution sequence and assigned participants to one of the two conditions (1:1 ratio).

Intervention: Mindfulness-Based Cognitive Therapy (MBCT) is a structured group intervention developed. The intervention consisted of eight weekly 2.5-hr sessions and one 3-hr silent session. The main aspects of the program; It included group meditation, cognitive-behavioral exercises, psycho-education, and daily homework. The intervention in our study closely followed the original manual, with several adaptations for the study group and purpose. First, psycho-education focused on the importance of recognizing personal feelings and the relationship between stress, postpartum blues, mother-infant attachment and breastfeeding symptoms, and stress management, stress, postpartum blues, mother-infant attachment and breastfeeding.

Control Condition: Postpartum mothers in the control condition were informed that they would receive MBCT after a waiting period of 2 months. Meanwhile, no psychological intervention was ofered.

Measures: The baseline questionnaire included questions about demographic, socioeconomic, obstetric, mood, and breastfeeding-specific information. Outcomes related to all stress, postpartum blues, mother-infant attachment, and breastfeeding were assessed at baseline and after therapy (on average, 2 months after baseline assessment).

Sample size calculation for the primary research question was performed based on a pilot study, which assessed pre- and post-measurement stres and depression levels in postpartum participating in a mindfulness program similar to MBCT, specifcally CALM Pregnancy as focused on training in formal mindfulness and informal mindfulness practices. The CALM Pregnancy program both involve eight weekly 2.5-hr sessions. Sessions included didactic presentations, group exercises, formal meditation practices, and leader-facilitated group inquiry and discussion. Formal practices included the body scan, mindful yoga, and sitting meditation. Informal mindfulness practices included mindfulness of everyday activities such as mindful eating and mindful walking. The intervention also incorporated the 3-min breathing space and cognitive approaches for developing alternative ways of responding to stress and anxiety symptoms. Given the similarities in the content, structure, and intensity of the two programs, the investigators used this pilot study for the sample size calculation. With a statistical power of 0.95 and an alpha of 0.05, 45 postpartum mothers patients were required per group (90 in total) to be able to detect diferences with an effect size of at least 0.50.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research,
* Over 18 years old,
* Participated in group sessions for 2,5 hours once a week for eight weeks,
* Mothers could read, write and speak Turkish.

Exclusion Criteria:

* Over 49 years old,
* The presence of serious cognitive, neurological, and psychiatric disorders that may preclude participation of postpartum mothers or require other treatment,
* Particularly psychotic complaints or a diagnosis of schizophrenia, neurological disorders including severe cognitive limitations,
* Substance use disorder, and acute suicidal thoughts or behaviors that may stress the mother,
* The presence of any congenital anomaly in the baby.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postpartum mothers
Enrollment: 90 (Actual)
Dates: Start 2022-04-02 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Stress evaluated using the Perceived Stress Scale | change from before implamentation patent and after 2 months of practice.
  The PSS-10, is a 14 items scale that was developed (Cohen et al., 1983) to assess perceived stress like the feelings and thoughts of one's life as uncontrollable, unpredictable, and overloaded over the last month with a five-point Likert (0: never, 4: very often) (e.g. "In the last month, how often have participants felt that things were going ones way?"). Scores on the PSS can range from 0 to 56 and higher scores indicate higher perceived stress. The scale was adapted to Turkish by Eskin and his colleagues (Eskin et al., 2013). During the adaptation to Turkish, the psychometric properties of the short-form of the 10-item and the 4-item scale, as well as the 14-item total scale, were tested. The internal consistency coefficients of the 14-item, 10-item, and 4-item forms of the scale were 0.84, 0.82, and 0.66; and test-retest reliability coefficients measured at one-month intervals were 0.87, 0.88, and 0.72, respectively. In this study, a ten-item short form of the scale was used.
Postpartum blues evaluated using the Edinburgh Postpartum Depression Scale | change from before implamentation patent and after 2 months of practice.
  This scale, which was developed to determine the risk of PPD, has been adapted to Turkish (Cox et al., 1987; Engindeniz et al., 1996). The scale consists of 10 items with 4 - point Likert-type responses. Each item is scored from 0-3, and the total score is obtained as the total of the item scores (min: 0 - max: 30). The cutoff point for the scale in Turkey has been calculated as 12/13 points (Engindeniz et al., 1996). In the current study, postpartum mothers with an EPDS score of ≥ 13 points were referred to the Psychiatry Department.
Mother-infant attachment evaluated using the Maternal Attachment Scale | change from before implamentation patent and after 2 months of practice.
  The MAS was developed by Müller (1994) and adapted to Turkish by Kavlak and Şirin (2009), was used to determine the level of the bond between mother and infant. The MAS includes 26 statements that people can use to express their feelings. Depending on the severity of the feelings of mothers against their babies, statements were calculated as 'Always=4 points, Frequently=3 points, Sometimes=2 points and Never=1 point'. An overall score was obtained from the sum of all items. High score indicates that maternal attachment is high. The scores obtained from the scale range from a minimum of 26 to a maximum of 104 points. The reliability coefficient of the MAS, which was adapted to Turkish by Kavlak and Şirin (2009), was found to be 0.77 in mothers with 1-month old newborn and 0.82 in mothers with 4-month old infant.
Breastfeeding blues evaluated using the Bristol Breastfeeding Assessment Scale | change from before implamentation patent and after 2 months of practice.
  The BBAS, which was developed by Ingram et al. (2014) and adapted into Turkish by Dolgun et al. (2018), was used in the study. The scale consists of 4 items (positioning, holding, sucking and swallowing) with 3 - point Likert-type responses. Each item is scored from 0-2 (0 poor, 1 moderate, 2 good), and the total score is obtained as the total of the item scores (min: 0 - max: 8). A high score indicates an effective breastfeeding or vice versa.

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey, Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided